CLINICAL TRIAL: NCT03634163
Title: Compassionate Communities Neighbourhood Program: Cluster Randomized Trial
Brief Title: Compassionate Communities Neighbourhood Program
Acronym: WECCC-NHB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Collaborators: Windsor-Essex Compassionate Care Community (Other); University of Windsor (Other); Hospice of Windsor and Essex County (Unknown); Erie St. Clair Local Health Integration Network (LHIN) (Other); Ontario Trillium Foundation (Other)
Responsible Party: Principal Investigator, Michelle Howard, Assistant Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 001-WECCC
Record Dates: First submitted 2018-07-05; First posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Chronic Disease; Aging
Keywords: disability
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: Cluster randomization with stepped wedge
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate (Experimental): Quality of Life Assessment plus facilitated implementation of neighbourhood exchange and personal care support
  Interventions: Behavioral: Neighbourhood exchange; Behavioral: Quality of Life Assessment
- Delayed (Active Comparator): Quality of Life Assessment
  Interventions: Behavioral: Quality of Life Assessment

INTERVENTIONS:
Behavioral: Neighbourhood exchange — Facilitated coaching support to identify needs and priorities and link with resources - personal, community, friend and family, or from professional service providers; plan and implement a personalized care pathway through community exchange
  Arms: Immediate
Behavioral: Quality of Life Assessment — Completion of baseline measures

SUMMARY:
This study will evaluate a Compassionate Communities-based intervention aimed at reducing social isolation by mobilizing individuals to act on their health and social needs individually, and in collaboration with fellow members of their community. The intervention program includes facilitated building of neighbourhood networks (member benefits include access to practical help, the opportunity to develop meaningful relationships, and community mobilization), and coaching support to work on individualized goal setting and more detailed navigation support and planning.

DETAILED DESCRIPTION:
The Compassionate Communities intervention is catalyzed by professional facilitators who visit communities with high concentrations of elderly and vulnerable residents, and recruit those who are interested in a project to identify their own health and social needs, assets and priorities; to collectively work to support each other in achieving these; and to implement a neighbourhood exchange to more easily match offers of help to people who need help. The mobilization work starts with the facilitator, who is employed by a community or social service organization, but increasingly draws on the energies of the mobilized initial participants as volunteers who conduct further community outreach in their community, attracting and mobilizing other residents, peers, and neighbouring resources in the work. Participants also plan and implement a broad range of activities identified by the residents as their priorities for neighbourhood building. Participants and their caregivers have the option of receiving more in-depth 1:1 coaching support to work on individualized goal setting, more detailed navigation support or advanced care planning following the sessions.

ELIGIBILITY:
Inclusion Criteria:

* Seniors (65 years of age and older)
* people with disabilities
* caregivers of seniors or people with disabilities
* residing in identified buildings/ neighbourhoods where the WECCC Compassionate Communities Neighbourhood program is being launched
* able to communicate in English or interpreter can be arranged

Exclusion Criteria:

* not able to communicate in English and interpreter cannot be arranged

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Perception of social disconnectedness | change from baseline at 7 months
  Social disconnectedness scale; 8-item validated scale (Cornwell and Waite, 2008), higher scores indicate greater social disconnectedness

SECONDARY OUTCOMES:
Perception of personal well-being | change from baseline at 7 months
  Assessed by Personal Well-Being Index (PWI); 8-item scale (Personal well-being index 5th edition, 2013). Higher scores indicate greater well-being
Perceived loneliness scale | change from baseline at 7 months
  Assessed by Perceived loneliness scale; 9-item validated scale (Cornwell and Waite, 2009). Higher scores indicated greater perceived isolation
Attainment of personal goals | Change from baseline at 7 months
  Assessed by Goal Attainment Scaling (GAS) instrument, measured on 5-point scale for each goal identified (Hurn et al, 2006), higher score indicates greater goal attainment
Health related quality of life | change from baseline at 7 months
  Assessed by Euroqol 5 dimension 5 level (5D-5L) scale; 5 levels of response for each of 5 items, score is converted to a single index, standardized to scale of 0 to 1, 1 being perfect health
Perceived provisions of social relationships | change from baseline at 7 months
  Social provisions scale; 10-item validated scale consisting of 5 subscales (Caron, 2013). The SPS 10 measures the perception of social support and consists of 10 items expressed as statements with responses coded on a 4-point scale from strongly disagree (= 1) to strongly agree (= 4). The total SPS-10 score is formed by the summation of raw scores, with high score indicating a higher degree of social provisions (maximum score of 40)
Number of emergency department visits | 7 months
  Number of emergency department visits measured from health administrative data
Number of hospital admissions | 7 months
  Number of hospital admissions measured from health administrative data

OTHER OUTCOMES:
Cost-effectiveness | 7 months
  Cost-effectiveness ratio measured as difference between groups in total health care utilization costs (measured from administrative data) divided by quality adjusted life years gained from the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Howard, PhD, Principal Investigator — McMaster University; Lisa Dolovich, PharmD, Principal Investigator — McMaster University; Kathryn Pfaff, PhD, Principal Investigator — University of Windsor; Merrick Zwarenstein, PhD, Principal Investigator — Western University; Denise Marshall, Principal Investigator — McMaster University; Ross Upshur, Principal Investigator — Sinai Health Systems; Carol Bennett, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Hospice of Windsor-Essex, Windsor, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided